CLINICAL TRIAL: NCT00936598
Title: Surgery for Endometrial Cancer: Biobehavioral Analysis of Sleep, Stress and Pain
Brief Title: Sleep and Endometrial Cancer
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Investigator-initiated termination of approval due to problems with recruitment.
Sponsor: University of Pittsburgh (Other)
Responsible Party: Principal Investigator, Dana Bovbjerg, Professor, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: PRO09040160; PCI-09-027 (Other: University of Pittsburgh Cancer Institute)
Record Dates: First submitted 2009-07-08; First posted 2009-07-10 (Estimated); Results first posted 2012-07-20 (Estimated); Last update posted 2014-04-24 (Estimated); Status verified 2014-04

CONDITIONS: Sleep; Endometrial Neoplasms; Pain
Keywords: Sleep; Endometrial Neoplasms; Pain
MeSH Terms: conditions — Endometrial Neoplasms; Pain | interventions — Zolpidem; Sugars

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- zolpidem (Experimental): Participants randomized to the zolpidem (intervention) group will receive the FDA approved dose of zolpidem, (10 mg for women <65; 5 mg for women > or = 65 years). For the purposes of this double-blind trial, zolpidem (e.g., Roxane Laboratories) pills will be placed without filler inside two-piece gelatin capsules (DBcaps, Capsugel) and packaged by the Investigational Drug Service (IDS) of the University of Pittsburgh Cancer Institute. During their presurgery visit (visit 1), participants will be provided with their capsule and instructed to take it by mouth immediately before bedtime the night before surgery.
  Interventions: Drug: zolpidem
- sugar pill (Placebo Comparator): Participants randomized to the sugar pill (control) group will receive placebo. For the purposes of this double-blind trial, placebo (sugar) pills will be placed without filler inside two-piece gelatin capsules (DBcaps, Capsugel) and packaged by the Investigational Drug Service (IDS) of the University of Pittsburgh Cancer Institute. During their presurgery visit (visit 1), participants will be provided with their capsule and instructed to take it by mouth immediately before bedtime the night before surgery.
  Interventions: Drug: sugar pill

INTERVENTIONS:
Drug: zolpidem — Participants will receive the FDA approved dose of zolpidem, (10 mg for women <65; 5 mg for women = or > 65 years) during their presurgery visit and will be instructed to take the single capsule by mouth immediately before bedtime the night before surgery.
  Other Names: Ambien
  Arms: zolpidem
Drug: sugar pill — Participants will receive placebo (sugar) pills during their presurgery visit and will be instructed to take the single capsule by mouth immediately before bedtime the night before surgery.
  Other Names: placebo
  Arms: sugar pill

SUMMARY:
This study proposes to test the hypothesis that zolpidem taken the night before major surgery for endometrial cancer will improve sleep efficiency and reduce post surgery pain, as well as reduce the need for analgesic medication.

DETAILED DESCRIPTION:
Despite continuing improvements in surgical procedures and ancillary care, post surgery pain continues to be a nearly universal patient experience following major operative procedures. Opioids provide considerable pain relief, but they have multiple adverse side effects and are not entirely effective. For cancer patients, uncontrolled postoperative pain can have a substantial negative effect on quality of life, can slow recovery, increase the likelihood of complications, and contribute to poorer postoperative outcomes. The identification of novel modifiable patient risk factors for post surgery pain that could become the target of presurgery interventions is thus an important goal. We will conduct a randomized, placebo-controlled, double-blind intervention trial design to evaluate the effects of an FDA approved hypnotic (zolpidem) on post surgery pain. Since presurgery psychological factors (e.g., heightened anxiety) are known to predict the severity of post surgical pain and may be associated with poor sleep, we will also assess psychological factors (with questionnaires) as well as sleep (using actigraphy) in order to determine their individual and combined impact on women's experiences of post surgery pain in this stressful clinical context. Aim 1: To determine the impact of zolpidem administered the night prior to endometrial cancer surgery on women's experiences of pain over the initial 7-10 day follow-up period after surgery using a double-blind placebo-controlled design (final n=128). Aim 2: To investigate psychological factors on the morning before surgery, as well as objective sleep variables on the night before surgery, as possible mediators of the beneficial effects of zolpidem on post surgery pain. Aim 3: To examine psychological factors, as well as sleep variables, assessed prior to the sleep intervention as possible moderators of the ameliorative effects of zolpidem on post surgery pain. The results of the proposed exploratory study would provide the preliminary data necessary for an R01 application to support more comprehensive investigations, including explorations of biological mechanisms underlying the preventative effects of better presurgery sleep on patients' experiences of post surgery pain.

ELIGIBILITY:
Inclusion Criteria:

* be women at least 18 years old
* have clinical indications of primary endometrioid adenocarcinoma of the endometrium
* be scheduled for staging surgery by laparotomy under standardized protocols
* have the ability to communicate in English sufficient for completion of study materials
* have no neuromuscular/ movement disorders (for actigraphy purposes)
* have no uncontrolled medical, sleep, endocrine or psychiatric illness (as determined by their attending physician as part of clinical care)
* have no ongoing use of medication known to affect sleep or wake function (e.g., hypnotics, benzodiazepines, antidepressants, anxiolytics, antipsychotics, decongestants, sedating antihistamines, beta blockers, corticosteroids)

Exclusion Criteria:

* have a history of previous or concomitant cancer
* have an estimated life expectancy of < 6 months
* will be admitted to the hospital prior to the day of surgery
* are unable to complete study measures
* are unable to provide meaningful informed consent

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2009-07; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dana H Bovbjerg, PhD, Principal Investigator — University of Pittsburgh
Locations (2):
- United States (2):
  - Magee-Womens Hospital of UPMC, Pittsburgh, Pennsylvania
  - UPMC Mercy, Pittsburgh, Pennsylvania

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment occurred between January 2010 and May 2010 at Magee Womens Hospital and Mercy Hospital. All participants who were recruited were assigned to one arm or the other.
Pre-assignment Details: One participant in the placebo group was found to be ineligible after consent before starting the study (before being provided with take home materials).
Groups:
- Zolpidem: Participants randomized to the Intervention group will receive the FDA approved dose of zolpidem, (10 mg for women <65; 5 mg for women > or = 65 years). For the purposes of this double-blind trial, zolpidem (e.g., Roxane Laboratories) and placebo (sugar) pills will be placed without filler inside two-piece gelatin capsules (DBcaps, Capsugel) and packaged by the Investigational Drug Service (IDS) of the University of Pittsburgh Cancer Institute.
- Sugar Pill: Participants in the Control group will receive placebo. For the purposes of this double-blind trial, zolpidem (e.g., Roxane Laboratories) and placebo (sugar) pills will be placed without filler inside two-piece gelatin capsules (DBcaps, Capsugel) and packaged by the Investigational Drug Service (IDS) of the University of Pittsburgh Cancer Institute.
Period: Overall Study
Arm/Group | Zolpidem | Sugar Pill
Started | 4 | 1
Completed | 2 | 1
Not Completed | 2 | 0
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Ineligible after consent | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Zolpidem | Sugar Pill | Total
Number analyzed (Participants) | 4 | 1 | 5
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 3 | 1 | 4
  >=65 years | 1 | 0 | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 53 (20.7) | 60 (0) | 54.4 (18.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 1 | 5
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 4 | 1 | 5

OUTCOME MEASURES:

1. Primary Outcome: Brief Pain Inventory (Short-form)
Description: Pain intensity and pain interference subscales from the Brief Pain Inventory (Short-form) (BPI) will be used to measure pain over the interval following surgery. Both subscales have a range of 0-10 with higher scores indicating worse outcomes (more intense pain and more pain interference).
Time Frame: at the clinical follow-up appointment approximately 7-10 days after surgery
Population: Due to limited enrollment in this study, and the small amount of data collected, we are unable to produce any significant results or conclusions.
Arm/Group | Zolpidem | Sugar Pill
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Pain Severity Visual Analogue Scale
Description: Pain severity will be assessed daily following surgery with a visual analogue scale (VAS) completed by participants each night before they go to bed (daily diary PM). VAS pain severity yields a score of 0 to 100, with 100 indicating pain "as bad as it could be."
Time Frame: each of the days following surgery until the clinical follow-up appointment
Population: as for outcome 1
Arm/Group | Zolpidem | Sugar Pill
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Daily Analgesic Medication Consumption (Morphine Equivalency)
Description: Analgesic medication consumption will be calculated (morphine equivalent daily dose (MEDD)) on a daily basis using data down loaded from the patient-controlled analgesia (PCA) pump supplemented by information from clinical charts and patient self report on the daily diary form. MEDD starts at zero and does not have an upper limit; higher daily doses indicate more analgesic medication consumption, and thus more pain.
Time Frame: daily from the day of surgery until the clinical follow-up appointment
Population: as for outcome 1
Arm/Group | Zolpidem | Sugar Pill
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Arm/Group | Zolpidem | Sugar Pill
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/1
Other Adverse Events (participants affected / at risk) | 0/4 | 0/1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No